CLINICAL TRIAL: NCT04560244
Title: Director of Shandong Cancer Hospital and Institute
Brief Title: A Trial of SHR1701 Combined With Radiotherapy for Metastatic Non-small Cell Lung Cancer Failure After First-line Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinming Yu, President of Shandong Cancer Hospital and Institute, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSCLC-2nd-IIT-SHR1701-RT
Record Dates: First submitted 2020-09-11; First posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: SHR1701,radiotherapy,NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — SHR-1701

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR 1701+radiotherapy (Experimental): SHR-1701 Simultaneously Combined with High Fractionation and Low-dose Radiotherapy
  Interventions: Drug: SHR1701

INTERVENTIONS:
Drug: SHR1701 — PD-L1 / TGF-β RII double antibody

SUMMARY:
This study is a single center, single arm, open study design. The main purpose of this study is to evaluate the tolerance and efficacy of SHR1701 with synchronous radiotherapy in patients with metastatic non-small cell lung cancer who have failed after systematic treatment. Large fraction radiotherapy is given to all lesions as much as possible, and low-dose radiotherapy is given to the lesions that cannot be tolerated or have no obvious benefit.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily participate in this study and sign informed consent.
* NSCLC in stage IV.
* No clear driven genes (including but not limited to EGFR、ALK、ROS1、cMET).
* Previously received more than 1 chemotherapy regimen and progressed/ recurred.
* At least one lesion is suitable for hypofraction radiotherapy.
* There is at least one measurable lesion.
* 18 to 75 years old
* ECOG 0-1
* The function of vital organs meets the following requirements. ANC ≥ 1.5×10^9/L, PLT≥100×10^9/L, Hb≥9g/dL, ALB≥3g/dL, TSH ≤ULN, Bilirubin ≤ 1 times ULN; ALT and AST ≤1.5 times ULN. AKP ≤ 2.5 times ULN. CREA ≤1.5 times ULN or CCr≥60mL/min#
* The estimated survival period is more than 3 months.
* Female Subjects of childbearing potential must have a negative serum pregnancy test within 72 hours before the first dose and must be willing to use very efficient barrier methods of contraception for the course of the study through 3 months after the last dose of study treatment

Exclusion Criteria:

The subjects had any history of autoimmune disease or active autoimmune disease.

* Subjects are using immunosuppressive agents, or systemic, or absorptive, local hormone therapy to achieve immunosuppression.It is still in use within 2 weeks of the entry.
* Subjects with severe allergic reactions to other monoclonal antibodies.
* The subjects had a central nervous system metastases of clinical symptoms.
* Central squamous cell lung carcinoma.
* Imaging (CT or MRI) shows that tumors invade large blood vessels or are indistinct with blood vessels.
* Imaging (CT or MRI) showed significant pulmonary vacuity or necrotic tumors,Borderline adenocarcinoma accompanied by a cavity can be considered after discussion with investigator.
* Failing to properly control the clinical symptoms or disease of the heart.
* Subjects had active infections.
* Subjects may receive other systemic antitumor therapy during the study period.
* Other clinical trials of drugs were used in the first four weeks of the first medication.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing adverse event (AE) | From the first administration of shr-1701 to 90 days after the last Administration
Number of participants experiencing serious adverse event (SAE) | From the first administration of shr-1701 to 90 days after the last Administration

SECONDARY OUTCOMES:
progression-free survival （PFS） | Up to approximately 24 months
Objective Response Rate （ORR） | Up to approximately 24 months
Disease control rate (DCR) | Up to approximately 24 months
Overall survival (OS) | Up to approximately 24 months

CONTACTS AND LOCATIONS:
Overall Officials: JinMing Yu, PhD, Principal Investigator — Shandong Cancer Hospital and Institute

IPD SHARING:
Plan to Share IPD: Undecided